CLINICAL TRIAL: NCT05510375
Title: Effect of Randomized Cocoa Supplementation on Inflammaging and Epigenetic Aging
Brief Title: Cocoa Supplementation, Inflammaging, and Epigenetic Aging
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Augusta University (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 1687423
Record Dates: First submitted 2021-09-15; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Aging; Inflammation; Cardiovascular Diseases
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases | interventions — Chocolate; Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cocoa extract + multivitamin (Active Comparator): Two capsules/day for 600 mg/day of cocoa flavanols One tablet/day of multivitamin
  Interventions: Dietary Supplement: Cocoa extract; Dietary Supplement: Multivitamin
- Cocoa extract + multivitamin placebo (Active Comparator): Two capsules/day for 600 mg/day of cocoa flavanols Multivitamin placebo
  Interventions: Dietary Supplement: Cocoa extract; Dietary Supplement: Multivitamin placebo
- Cocoa extract placebo + multivitamin (Active Comparator): Cocoa extract placebo One tablet/day of multivitamin
  Interventions: Dietary Supplement: Multivitamin; Dietary Supplement: Cocoa extract placebo
- Cocoa extract placebo + multivitamin placebo (Placebo Comparator): Cocoa extract placebo Multivitamin placebo
  Interventions: Dietary Supplement: Cocoa extract placebo; Dietary Supplement: Multivitamin placebo

INTERVENTIONS:
Dietary Supplement: Cocoa extract — 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin, and 50 mg theobromine
  Arms: Cocoa extract + multivitamin; Cocoa extract + multivitamin placebo
Dietary Supplement: Multivitamin — Multivitamin
  Arms: Cocoa extract + multivitamin; Cocoa extract placebo + multivitamin
Dietary Supplement: Cocoa extract placebo — Cocoa extract placebo
  Arms: Cocoa extract placebo + multivitamin; Cocoa extract placebo + multivitamin placebo
Dietary Supplement: Multivitamin placebo — Multivitamin placebo
  Arms: Cocoa extract + multivitamin placebo; Cocoa extract placebo + multivitamin placebo

SUMMARY:
The COcoa Supplement and Multivitamin Outcomes Study (COSMOS; NCT02422745) is a randomized clinical trial of cocoa extract supplement (containing a total of 500 mg/d flavanols, including 80 mg. (-)-epicatechins), and a standard multivitamin supplement to reduce the risk of cardiovascular disease and cancer among men aged 60 years and older and women aged 65 years and older. This ancillary study is being conducted among participants in COSMOS and will examine whether the cocoa extract supplement or the multivitamin supplement has an anti-aging effect (epigenetic aging and inflammaging) and examining these findings in the context of CVD risk factors and outcomes.

ELIGIBILITY:
Participants in COSMOS (NCT02422745) who meet the following criteria are eligible to participate in this ancillary study:

Inclusion Criteria:

* Provided blood samples at baseline, Year 1, and Year 2 of follow-up.
* Opted to use EMSI for longitudinal blood collections, during which seated BPs were additionally measured.

Exclusion Criteria:

• Did not collect blood samples at baseline, Year 1, or Year 2 of follow-up.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21442 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Epigenetic age acceleration | 2 years
  A cumulative epigenetic aging index (DNAm age) that predicts DNAm age will be calculated. The residual from regressing DNAm age on chronological age provides a measure of epigenetic age acceleration.
Inflammaging | 2 years
  An index constructed using several inflammation markers reflecting inflammaging.

SECONDARY OUTCOMES:
Blood pressure | 2 years
  Systolic and diastolic blood pressure in mmHg.
Body mass index | 2 years
  Body mass index in kg/m2 will be calculated using height and weight
Pulse wave velocity | 2 years
  Pulse wave velocity in m/s from the carotid to the femoral artery will be measured.